CLINICAL TRIAL: NCT06484608
Title: Comparison of Isotonic Versus Hypotonic Fluids in Neonates Receiving Maintenance Fluid Therapy Post-Surgery: A Randomized Controlled Trial
Brief Title: Comparison of Isotonic Versus Hypotonic Fluids in Neonates for Maintenance Fluid Therapy After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Mehak Fatima, Mehak Fatima, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RawalpindiMU
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hyponatremia; Hypernatremia; Postoperative Care in Neonates; Edema
Keywords: isotonic saline, hypotonic saline, neonates, maintenance fluid therapy, surgery, hyponatremia
MeSH Terms: conditions — Hyponatremia; Hypernatremia; Edema | interventions — Sodium Chloride; Glucose

STUDY DESIGN:
Intervention Model Description: In this study, participants (neonates post-surgery) are randomly assigned to one of two groups, with each group receiving a different type of intervention (isotonic or hypotonic fluids). The parallel assignment model means that all participants in each group receive the same intervention throughout the study period, and the outcomes of these groups are compared to evaluate the effectiveness and safety of the interventions.
Who Masked: Participant
Masking Description: In this study, masking is implemented at the participant level. This means that the neonates (participants) and their caregivers are unaware of whether the neonate is receiving isotonic or hypotonic fluids. However, the clinical staff administering the fluids and assessing outcomes are not blinded to the intervention group. This approach helps reduce bias in the perception and reporting of outcomes by those caring for the neonates while ensuring accurate administration and monitoring by the healthcare providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isotonic Fluid Group (Experimental): Neonates in this group will receive isotonic/normal saline with 5% dextrose in 0.9% saline as their maintenance fluid therapy post-surgery. This intervention aims to maintain serum sodium levels and reduce the risk of hyponatremia and other complications.
  Interventions: Drug: Isotonic Saline with Dextrose
- Hypotonic Fluid Group (Active Comparator): Neonates in this group will receive hypotonic saline with 5% dextrose in 0.45% saline as their maintenance fluid therapy post-surgery. This intervention is being compared to isotonic fluid therapy to evaluate its effectiveness and safety in maintaining electrolyte balance and preventing hypernatremia and edema.
  Interventions: Drug: Isotonic Saline with Dextrose

INTERVENTIONS:
Drug: Isotonic Saline with Dextrose — This clinical trial involves two interventions for maintaining fluid therapy in neonates post-surgery. The first intervention, isotonic saline with dextrose, involves administering 0.9% saline solution combined with 5% dextrose. This isotonic solution aims to maintain serum sodium levels within the normal range and minimize the risk of hyponatremia and hypernatremia in postoperative neonates. The second intervention, hypotonic saline with dextrose, involves administering 0.45% saline solution combined with 5% dextrose. This hypotonic solution is being compared to the isotonic solution to evaluate its effectiveness in maintaining electrolyte balance.
  Other Names: Hypotonic Saline with Dextrose

SUMMARY:
The goal of this clinical trial is to determine if isotonic or hypotonic fluids are more effective in maintaining serum sodium levels in neonates undergoing maintenance fluid therapy post-surgery. The main questions it aims to answer are:

Does isotonic fluid therapy reduce the risk of hyponatremia compared to hypotonic fluid therapy? Does hypotonic fluid therapy lead to fewer cases of hypernatremia compared to isotonic fluid therapy? Researchers will compare neonates receiving isotonic fluids (Group I: isotonic/normal saline with 5% dextrose in 0.9% saline) to those receiving hypotonic fluids (Group H: hypotonic saline with 5% dextrose in 0.45% saline) to see if there are significant differences in serum sodium levels and associated complications.

Participants will:

Be randomly assigned to receive either isotonic or hypotonic fluids. Have blood samples taken before and after surgery to assess serum sodium levels.

Be monitored for 24 hours post-surgery to observe any complications such as hyponatremia, hypernatremia, or edema.

This study enrolled 84 neonates admitted to the neonatal intensive care unit following surgery, and data analysis was conducted using SPSS software version 25.0.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to determine the most appropriate type of maintenance fluid (isotonic versus hypotonic) for neonates following surgery. The study enrolled 84 neonates, aged 1-28 days, who were admitted to the neonatal intensive care unit at Holy Family Hospital Rawalpindi from January 2023 to December 2023.

Neonates were randomly assigned into two groups:

Group I: Received isotonic/normal saline with 5% dextrose in 0.9% saline. Group H: Received hypotonic saline with 5% dextrose in 0.45% saline. Blood samples were collected before surgery and 24 hours post-surgery to measure serum sodium levels. The main outcome measures were the incidence of hyponatremia (serum sodium level <135 mEq/L) and hypernatremia (serum sodium level >145 mEq/L). Secondary outcomes included other complications such as edema.

The results indicated that:

Hyponatremia occurred in 2 (4.8%) cases in the isotonic group and 11 (26.2%) cases in the hypotonic group.

Hypernatremia was observed in 9 (21.4%) cases in the isotonic group and none in the hypotonic group.

Edema was noted in 1 (2.4%) neonate in the isotonic group and 9 (21.4%) neonates in the hypotonic group.

The study concluded that isotonic saline is more effective in maintaining normal serum sodium levels and reducing the risk of hyponatremia and other complications compared to hypotonic saline in neonates post-surgery. Further research with larger sample sizes and additional electrolyte considerations is recommended to improve outcomes and reduce morbidity and mortality in this population.

ELIGIBILITY:
Inclusion Criteria:

* Neonates aged 1-28 days. Admitted to the neonatal intensive care unit (NICU) at Holy Family Hospital Rawalpindi.

Scheduled for surgery requiring maintenance fluid therapy postoperatively. Parental or guardian consent obtained.

Exclusion Criteria:

* Neonates with pre-existing electrolyte imbalances or metabolic disorders. Neonates with congenital heart disease or renal impairment. Neonates on diuretics or other medications affecting fluid balance. Neonates with a history of intrauterine growth restriction (IUGR). Neonates with major congenital anomalies. Lack of parental or guardian consent.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Hyponatremia and Hypernatremia | Before surgery (baseline measurement) 24 hours post-surgery
  This outcome measures the incidence of hyponatremia (serum sodium level <135 mEq/L) and hypernatremia (serum sodium level >145 mEq/L) in neonates receiving either isotonic or hypotonic saline with dextrose as maintenance fluid therapy post-surgery

SECONDARY OUTCOMES:
Incidence of Edema | Before surgery (baseline measurement) 24 hours post-surgery
  This outcome measures the incidence of edema in neonates receiving either isotonic or hypotonic saline with dextrose as maintenance fluid therapy post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mehak Fatima, MBBS, Principal Investigator — RMU
Locations (1):
- Mehak Fatima, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The plan for sharing individual participant data (IPD) is currently undecided. We recognize the importance of data sharing to advance scientific knowledge and improve clinical practices. We are considering several factors, including patient privacy, ethical considerations, and the logistics of data management, to make an informed decision. If a decision to share data is made in the future, we will outline the conditions under which the data will be shared, the type of data to be shared, and the means by which interested researchers can access the data. Any IPD sharing will be conducted in accordance with applicable regulations and ethical guidelines to ensure the protection of participant confidentiality and data integrity.